CLINICAL TRIAL: NCT01537185
Title: A Phase 1 Randomized, Double-Blind, Dose-Escalation Study to Assess the Safety, Tolerability and Immunogenicity of Inactivated Streptococcus Pneumoniae Whole Cell Vaccine Formulated With Alum (SPWCV+Alum) in Healthy Adults
Brief Title: Phase I Safety Trial of Streptococcus Pneumoniae Whole Cell Vaccine (SPWCV) + Alum in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH Vaccine Solutions (Other)
Responsible Party: Sponsor
Organization: PATH (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAC 002
Record Dates: First submitted 2012-02-07; First posted 2012-02-23 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2012-02

CONDITIONS: Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 SPWCV+Alum 100 mcg (Experimental): each individual receiving 3 vaccinations of same dose 28 days apart
  Interventions: Biological: SPWCV+Alum 100 mcg
- Cohort 2 SPWCV+Alum 300 mcg (Experimental): each individual receiving 3 vaccinations of same dose 28 days apart
  Interventions: Biological: SPWCV+Alum 300 mcg
- Cohort 3 SPWCV+Alum 600 mcg (Experimental): each individual receiving 3 vaccinations of same dose 28 days apart
  Interventions: Biological: SPWCV+Alum 600 mcg
- Normal Saline Injection (Placebo Comparator): placebo group within each cohort receive 3 injections of normal saline 28 days apart
  normal saline injection: 3 cohorts of normal saline injection
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — 3 cohorts of normal saline injection
  Arms: Normal Saline Injection
Biological: SPWCV+Alum 100 mcg — 3 injections 28 days apart
  Arms: Cohort 1 SPWCV+Alum 100 mcg
Biological: SPWCV+Alum 600 mcg — 3 injections 28 days apart
  Arms: Cohort 3 SPWCV+Alum 600 mcg
Biological: SPWCV+Alum 300 mcg — 3 injections 28 days apart
  Arms: Cohort 2 SPWCV+Alum 300 mcg

SUMMARY:
The purpose of this study is to determine if a Streptococcus pneumoniae Whole Cell Vaccine (SPWCV) given with alum is safe and well tolerated by healthy adults.

ELIGIBILITY:
Inclusion Criteria, Healthy adults:

* If female, not breastfeeding, not pregnant, not planning pregnancy during study period), and willing to consistently use an adequate method of contraception and have repeated pregnancy tests.
* In good health with normal laboratory results
* Willing to comply with study restrictions, study schedule, and can be reliably contacted

Exclusion Criteria:

* Currently consumes alcohol in excess of 2 drinks per day for men or 1 drink per day for women.
* current use or likely requirement for medications with potential for liver injury or effect immune system
* History of event or condition such as anaphylaxis, severe allergic reactions, serious reactions to any vaccines, or other events that might increase risk of reaction to an investigational disease
* History of diabetes, cancer, autoimmune or immunosuppressive disease or chronic such as HIV, Hepatitis B or C

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Royce Morrison, M.D., Principal Investigator — Comprehensive Clinical Development
Locations (1):
- Comprehensive Clinical Development, Tacoma, Washington, United States

REFERENCES:
- [Derived] Keech CA, Morrison R, Anderson P, Tate A, Flores J, Goldblatt D, Briles D, Hural J, Malley R, Alderson MR. A Phase 1 Randomized, Placebo-controlled, Observer-blinded Trial to Evaluate the Safety and Immunogenicity of Inactivated Streptococcus pneumoniae Whole-cell Vaccine in Adults. Pediatr Infect Dis J. 2020 Apr;39(4):345-351. doi: 10.1097/INF.0000000000002567. PMID 31895881
- [Derived] Campo JJ, Le TQ, Pablo JV, Hung C, Teng AA, Tettelin H, Tate A, Hanage WP, Alderson MR, Liang X, Malley R, Lipsitch M, Croucher NJ. Panproteome-wide analysis of antibody responses to whole cell pneumococcal vaccination. Elife. 2018 Dec 28;7:e37015. doi: 10.7554/eLife.37015. PMID 30592459

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 2 SPWCV+Alum 300 mcg; Cohort 3 SPWVC+Alum 600 mcg: each individual receiving 3 vaccinations of the same dose 28 days apart
Period: Overall Study
Arm/Group | Cohort 1 SPWCV+Alum 100 mcg | Normal Saline Injection | Cohort 2 SPWCV+Alum 300 mcg | Cohort 3 SPWVC+Alum 600 mcg
Started | 10 | 12 | 10 | 10
Completed | 7 | 6 | 4 | 8
Not Completed | 3 | 6 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 SPWCV+Alum 100 mcg | Normal Saline Injection | Cohort 2 SPWCV+Alum 300 mcg | Cohort 3 SPWCV+Alum 600 mcg | Total
Number analyzed (Participants) | 10 | 12 | 10 | 10 | 42
Age, Continuous [Mean (Full Range); unit: years] | 28.9 [19 to 40] | 28.5 [18 to 40] | 25.2 [18 to 34] | 29.9 [21 to 40] | 28.1 [18 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 4 | 7 | 22
  Male | 7 | 4 | 6 | 3 | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 10 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Unsolicited Adverse Event Reports
Description: Safety and Tolerability assessed by cohort and product received measured by:
  •Number of unsolicited AEs within four weeks after each vaccination
Time Frame: within 1 week (0-7 days) following each vaccinations
Measure: Number; unit: participants
Arm/Group | Cohort 1 SPWCV+Alum 100 mcg | Normal Saline Injection | Cohort 2 SPWCV+Alum 300 mcg | Cohort 3 SPWVC+Alum 600 mcg
Number analyzed (Participants) | 10 | 12 | 10 | 10
participants | 7 | 6 | 5 | 6

2. Secondary Outcome: Immunogenicity Determined by the Number of Subjects With >4x Increase in Anti IgG
Description: • Determination of a humoral immune response to whole cell antigen as determined by ELISA of sera collected on Day 0, 28, 56, and 84.
Time Frame: 28, 56 and 84 days following initial vaccination
Population: only subjects with both baseline and day 84 samples were included in the analysis.
Measure: Number; unit: participants
Groups:
- Cohort 3 SPWVC+Alum 600 mcg: each individual receiving 3 vaccinations of same dose 28 days apart
Arm/Group | Cohort 1 SPWCV+Alum 100 mcg | Normal Saline Injection | Cohort 2 SPWCV+Alum 300 mcg | Cohort 3 SPWVC+Alum 600 mcg
Number analyzed (Participants) | 9 | 9 | 5 | 9
participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Cohort 1 SPWCV+Alum 100 mcg | Normal Saline Injection | Cohort 2 SPWCV+Alum 300 mcg | Cohort 3 SPWCV+Alum 600 mcg
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/12 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 6/12 | 5/10 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 SPWCV+Alum 100 mcg (N=10) | Normal Saline Injection (N=12) | Cohort 2 SPWCV+Alum 300 mcg (N=10) | Cohort 3 SPWCV+Alum 600 mcg (N=10)
ruptured ectopic pregnancy with hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 SPWCV+Alum 100 mcg (N=10) | Normal Saline Injection (N=12) | Cohort 2 SPWCV+Alum 300 mcg (N=10) | Cohort 3 SPWCV+Alum 600 mcg (N=10)
neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
viral infection (Infections and infestations) | 0 | 1 | 0 | 0
viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
haemoglobin decreased (Investigations) | 0 | 2 | 1 | 2
platelet count decreased (Investigations) | 1 | 0 | 0 | 0
hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 2
dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Endodontic Procedure (Surgical and medical procedures) | 0 | 0 | 0 | 1
injection site pain (General disorders) | 0 | 0 | 2 | 1
irritability (General disorders) | 0 | 0 | 0 | 1
tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less